CLINICAL TRIAL: NCT01152359
Title: Considering Patient Diet Preference to Optimize Weight Loss
Brief Title: Considering Patient Diet Preferences to Optimize Weight Loss
Acronym: DietChoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 09-381
Record Dates: First submitted 2010-06-14; First posted 2010-06-29 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: obesity; diet, low carbohydrate; diet, fat-restricted; food preferences; quality of life; patient compliance
MeSH Terms: conditions — Obesity; Food Preferences; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Participants are allowed to choose between a low-carbohydrate or a low-fat diet for weight loss after receiving information about these diets and their food preferences (Choice arm). Then they receive counseling on their chosen diet in a small group format. The low-carbohydrate diet limits carbohydrate intake to 20-40 grams/day initially. The low-fat diet restricts saturated fat to below 30% of daily calories and has a 500-1000 calorie deficit. Group sessions are every 2 weeks for 24 weeks then alternate with telephone calls every 2 weeks for 24 weeks. Phone calls focus on goal setting to maximize weight loss. Participants also receive counseling on behavioral techniques and physical activity. Participants in this arm have the option to switch diets at 12 weeks.
  Interventions: Behavioral: Choice
- Arm 2 (Active Comparator): Participants are randomly assigned to (rather than getting to choose, as in the experimental arm) a low-carbohydrate or a low-fat diet for weight loss (Control arm). Then they receive counseling on their chosen diet in a small group format. The low-carbohydrate diet limits carbohydrate intake to 20-40 grams/day initially. The low-fat diet restricts saturated fat to below 30% of daily calories and has a 500-1000 calorie deficit. Group sessions are every 2 weeks for 24 weeks then alternate with telephone calls every 2 weeks for 24 weeks. Phone calls focus on goal setting to maximize weight loss. Participants also receive counseling on behavioral techniques and physical activity. Participants in this arm do not have the option to switch diets at 12 weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Choice — Participants are allowed to choose between a low-carbohydrate or a low-fat diet for weight loss after receiving information about these diets and their food preferences (Choice arm). Then they receive counseling on their chosen diet in a small group format. The low-carbohydrate diet limits carbohydrate intake to 20-40 grams/day initially. The low-fat diet restricts saturated fat to below 30% of daily calories and has a 500-1000 calorie deficit. Group sessions are every 2 weeks for 24 weeks then alternate with telephone calls every 2 weeks for 24 weeks. Phone calls focus on goal setting to maximize weight loss. Participants also receive counseling on behavioral techniques and physical activity. Participants in this arm have the option to switch diets at 12 weeks.
  Arms: Arm 1
Behavioral: Control — Participants are randomly assigned to (rather than getting to choose, as in the experimental arm) a low-carbohydrate or a low-fat diet for weight loss (Control arm). Then they receive counseling on their chosen diet in a small group format. The low-carbohydrate diet limits carbohydrate intake to 20-40 grams/day initially. The low-fat diet restricts saturated fat to below 30% of daily calories and has a 500-1000 calorie deficit. Group sessions are every 2 weeks for 24 weeks then alternate with telephone calls every 2 weeks for 24 weeks. Phone calls focus on goal setting to maximize weight loss. Participants also receive counseling on behavioral techniques and physical activity. Participants in this arm do not have the option to switch diets at 12 weeks.
  Arms: Arm 2

SUMMARY:
Obesity is increasingly common and can lead to decreased quality of life, increased medical and psychiatric illness, high health care costs, and early mortality. The problem of obesity is as great in veterans as it is in the general public. Adherence to dietary therapy for obesity is often inadequate, possibly because patients' food preferences are not considered during dietary counseling. Allowing patients to choose a diet based on their food preferences may increase their motivation to adhere to diet counseling. This, in turn, could enhance their weight loss success and, ultimately, reduce the many health complications and costs of obesity. The proposed study will examine whether assessing a person's food preferences, and then allowing the person to choose from two commonly prescribed diets, results in greater weight loss success.

DETAILED DESCRIPTION:
The prevalence of obesity (body mass index [BMI] 30 kg/m2) in US adults has skyrocketed over the past 30 years, and is currently as high or higher in veterans as it is in non-veterans. Thus, identifying effective strategies for treating obesity is both a public health and a VA priority. A variety of diet approaches have proven successful in achieving moderate weight loss in many individuals. Yet, most diet interventions fail to achieve meaningful weight loss in more than a few individuals. This failure likely results from inadequate adherence to the diet.

It is widely felt, but not empirically shown, that targeting the diet to an individual's food preferences will enhance adherence, thereby improving weight loss outcomes. This study will test the commonly proposed assumption that helping patients choose a diet based on their dietary preferences will increase weight loss success relative to assigning or recommending one diet.

The proposed study is a 2-arm randomized controlled trial involving 216 outpatients from Durham VA Medical Center. Participants must be obese (BMI 30 kg/m) VAMC outpatients without unstable health issues. Participants in the experimental arm (Choice) will select from two of the most widely studied diets for weight loss, either a low-carbohydrate, calorie-unrestricted diet (LCD) or a low-fat, reduced-calorie diet (LFD). This choice will be informed by results from a validated food preference questionnaire and a discussion of available diet options with trained personnel. As may occur in the clinical setting, the Choice participants will also have the opportunity to switch to the other diet after 3 months if unsuccessful or dissatisfied with their primary selection. The Choice intervention is designed to enhance the three psychological needs of a person according to self-determination theory (SDT): competence, relatedness, and, in particular, autonomy. This should maximize intrinsic motivation, thereby improving adherence to diet recommendations and increasing weight loss. Participants in the Control arm will be randomly assigned to follow one of the two diets for the duration of follow-up.

All participants will receive diet-appropriate counseling in small group meetings every 2 weeks for 24 weeks, then monthly for another 24 weeks. All participants will also receive brief telephone counseling involving individual goal setting and problem solving halfway through each month in the latter 24 weeks. The primary outcome is weight change from baseline to 48 weeks. Secondary outcomes include adherence to diet by food frequency questionnaire and obesity-specific health-related quality of life. Exploratory analyses will examine whether the impact of choice versus lack of choice on weight loss is moderated by individual differences in the SDT constructs of autonomy orientation, competence, and relatedness.

If assisting patients to choose their diet enhances adherence and increases weight loss, the results will support the provision of diet options to veterans and non-veterans alike, and bring us one step closer to remediating the obesity epidemic faced by the VA and other healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30 or greater
* Stable health
* Desire to lose weight
* Agrees to attend regular visits
* Access to telephone and reliable transportation
* Has a Veterans Affairs Medical Center (VAMC) provider

Exclusion Criteria:

* Certain chronic or unstable disease (kidney or liver disease, type 1 diabetes, hemoglobin A1c 12% or more, insulin use, unstable heart disease, transplant recipient, blood pressure 160/100 or greater, fasting blood triglycerides 600 or greater, LDL cholesterol 190 or greater)
* Pregnancy, breastfeeding, lack of birth control
* Active dementia, psychiatric illness, or substance abuse (past year)
* Weight loss therapy in previous month
* Pacemaker or defibrillator
* Enrolled in another study that might affect measurements
* Previously in study of low-carbohydrate or low-fat diet for weight loss
* Unable to complete all study measures

Max Age: 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S. Yancy, MD MHS, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Background] McVay MA, Yancy WS Jr, Vijan S, Van Scoyoc L, Neelon B, Voils CI, Maciejewski ML. Obesity-related health status changes and weight-loss treatment utilization. Am J Prev Med. 2014 May;46(5):465-72. doi: 10.1016/j.amepre.2013.11.018. PMID 24745636
- [Background] Yancy WS. Peer Support Significantly Improves Compliance in Veterans with Diabetes. U. S. Medicine. 2012 Nov 20.
- [Result] Yancy WS Jr, McVay MA, Brinkworth GD. Adherence to diets for weight loss. JAMA. 2013 Dec 25;310(24):2676. doi: 10.1001/jama.2013.282639. No abstract available. PMID 24368474
- [Result] McVay MA, Jeffreys AS, King HA, Olsen MK, Voils CI, Yancy WS Jr. The relationship between pretreatment dietary composition and weight loss during a randomised trial of different diet approaches. J Hum Nutr Diet. 2015 Feb;28 Suppl 2:16-23. doi: 10.1111/jhn.12188. Epub 2013 Nov 20. PMID 24251378
- [Result] McVay MA, Voils CI, Coffman CJ, Geiselman PJ, Kolotkin RL, Mayer SB, Smith VA, Gaillard L, Turner MJ, Yancy WS Jr. Factors associated with choice of a low-fat or low-carbohydrate diet during a behavioral weight loss intervention. Appetite. 2014 Dec;83:117-124. doi: 10.1016/j.appet.2014.08.023. Epub 2014 Aug 19. PMID 25149197
- [Result] Yancy WS Jr, Coffman CJ, Geiselman PJ, Kolotkin RL, Almirall D, Oddone EZ, Mayer SB, Gaillard LA, Turner M, Smith VA, Voils CI. Considering patient diet preference to optimize weight loss: design considerations of a randomized trial investigating the impact of choice. Contemp Clin Trials. 2013 May;35(1):106-16. doi: 10.1016/j.cct.2013.03.002. Epub 2013 Mar 16. PMID 23506974
- [Result] Yancy WS Jr, Mayer SB, Coffman CJ, Smith VA, Kolotkin RL, Geiselman PJ, McVay MA, Oddone EZ, Voils CI. Effect of Allowing Choice of Diet on Weight Loss: A Randomized Trial. Ann Intern Med. 2015 Jun 16;162(12):805-14. doi: 10.7326/M14-2358. PMID 26075751
- [Result] Yancy WS Jr, McVay MA, Voils CI. Effect of allowing choice of diet on weight loss--in response. Ann Intern Med. 2015 Nov 17;163(10):805-6. doi: 10.7326/L15-5159. No abstract available. PMID 26571246
- [Result] McVay MA, Voils CI, Geiselman PJ, Smith VA, Coffman CJ, Mayer S, Yancy WS Jr. Food preferences and weight change during low-fat and low-carbohydrate diets. Appetite. 2016 Aug 1;103:336-343. doi: 10.1016/j.appet.2016.04.035. Epub 2016 Apr 29. PMID 27133551

RESULTS

PARTICIPANT FLOW:
Groups:
- Choice Arm: Upon starting the study, participants are able to make an informed choice between a low-carbohydrate or a low-fat diet for weight loss after receiving information about these diets and about their food preferences as assessed by a questionnaire. Then participants will receive counseling regarding their chosen diet in a small group format. Sessions will take place every 2 weeks for 24 weeks then group sessions will alternate with telephone calls every 2 weeks for 24 weeks. Phone calls will focus on goal setting to maximize weight loss. In addition to counseling on diet during group sessions and phone calls, participants will receive counseling on behavioral techniques and physical activity.
- Control Arm: Upon starting the study, participants are randomly assigned to a low-carbohydrate or a low-fat diet for weight loss. Then participants will receive counseling regarding their chosen diet in a small group format. Sessions will take place every 2 weeks for 24 weeks then group sessions will alternate with telephone calls every 2 weeks for 24 weeks. Phone calls will focus on goal setting to maximize weight loss. In addition to counseling on diet during group sessions and phone calls, participants will receive counseling on behavioral techniques and physical activity.
Period: Overall Study
Arm/Group | Choice Arm | Control Arm
Started | 105 | 102
Completed | 81 | 80
Not Completed | 24 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Choice Arm | Control Arm | Total
Number analyzed (Participants) | 105 | 102 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 55 (10) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 77 | 75 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 61 | 106
  White | 54 | 39 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 105 | 102 | 207

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline to 48 Weeks
Time Frame: Baseline, 48 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of weight change
Arm/Group | Choice Arm | Control Arm
Number analyzed (Participants) | 105 | 102
percentage of weight change | -4.2 [-5.0 to -3.4] | -5.3 [-6.1 to -4.4]
Statistical Analysis 1: Comparison: Choice Arm vs Control Arm; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.8 to 2.9]

2. Secondary Outcome: Diet Adherence as Measured by Block Food-frequency Questionnaire (Absolute Percentage Deviation From the Goal Macronutrient Intake--<30% Fat for Low-fat Diet or <10% Carbohydrate for Low-carbohydrate Diet)
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of deviation from goal
Arm/Group | Choice Arm | Control Arm
Number analyzed (Participants) | 105 | 102
percentage of deviation from goal | 9.4 [6.6 to 12.3] | 10.3 [7.5 to 13.1]
Statistical Analysis 1: Comparison: Choice Arm vs Control Arm; Test type: Superiority; p = 0.66, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-4.9 to 3.1]

3. Secondary Outcome: Change in Obesity-specific Health-related Quality of Life as Measured by Impact Of Weight On Quality Of Life-Lite (IWQOL-Lite) Questionnaire From Baseline to 48 Weeks
Description: change in obesity-specific health-related quality of life as measured by Impact Of Weight On Quality Of Life-Lite (IWQOL-Lite) Questionnaire total score from baseline to 48 weeks Minimum 0 Maximum 100 Higher score means better
Time Frame: Baseline, 48 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Choice Arm | Control Arm
Number analyzed (Participants) | 105 | 102
score on a scale | 10.5 [8.0 to 12.9] | 11.2 [8.8 to 13.6]
Statistical Analysis 1: Comparison: Choice Arm vs Control Arm; Test type: Superiority; p = 0.65, Mixed Models Analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.1 to 2.6]

ADVERSE EVENTS:
Arm/Group | Choice Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 4/105 | 4/102
Other Adverse Events (participants affected / at risk) | 17/105 | 10/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Choice Arm (N=105) | Control Arm (N=102)
CHF (Cardiac disorders) | 1 (1) | 0 (0)
hip surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
spine surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gallbladder surgery (Hepatobiliary disorders) | 0 (0) | 1 (1)
finger infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
snake bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Choice Arm (N=105) | Control Arm (N=102)
Elevated blood pressure (Vascular disorders) | 8 (9) | 3 (3)
broken hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
lumps in hand (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
presyncope (Vascular disorders) | 1 (1) | 2 (2)
angioedema (Immune system disorders) | 1 (1) | 0 (0)
inner ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypoglcyemia (Endocrine disorders) | 1 (1) | 0 (0)
kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
motor vehicle collision (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (3)
dysphonia/vocal cord disorder (Nervous system disorders) | 0 (0) | 1 (1)
carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes